CLINICAL TRIAL: NCT00688922
Title: Pravastatin for Acute Myocardial Infarction With Minimally to Mildly Increased Levels of Serum Cholesterol Study That Evaluates the Effects of Pravastatin for Acute Myocardial Infarction With LDL-Cholesterol Levels of 70-129 mg/dl
Brief Title: Pravastatin for Acute Myocardial Infarction With Minimally to Mildly Increased Levels of Serum Cholesterol Study
Acronym: PRACTIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka Acute Coronary Insufficiency Study Group (Other)
Responsible Party: Hiroshi Sato, Osaka University Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRACTIC080703
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pravastatin — Take an initial dose of pravastatin to start as 10mg/day, which is the recommended initial dose by Health, Labour and Welfare Ministry of Japan, and a diet counseling.

SUMMARY:
The purpose of the Study is to determine whether early treatment with pravastatin can reduce adverse cardiac events in patients with acute myocardial infarction and minimally to mildly elevated serum Low Density Lipoprotein -Cholesterol (LDL-C) levels.

DETAILED DESCRIPTION:
The investigators previously reported the beneficial effect of early use of low-dose pravastatin on major adverse cardiac events in patients with acute myocardial infarction and mild to moderate hypercholesterolemia in the OACIS-LIPID Study. The PRACTIC study is designed as the OACIS-LIPID II trial to determine whether early treatment with pravastatin can reduce adverse cardiac events in patients with acute myocardial infarction and minimally to mildly elevated serum Low Density Lipoprotein -Cholesterol (LDL-C) levels.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of 2 of the following 3 criteria:

   1. a clinical history of central chest oppression, pain, or tightness lasting for ≥30 minutes
   2. typical electrocardiographic changes (i.e., ST-segment elevation of >0.1 mV in ≥1 limb or 2 precordial leads, ST-segment depression >0.1 mV in ≥2 leads, abnormal Q waves, or T-wave inversion in ≥2 leads)
   3. an increase in the serum creatine kinase levels to >2 times the normal laboratory value.
2. the serum level of LDL-C is ≥70 and 130> mg/dl in the first blood examination soon after admission

Exclusion Criteria:

1. concurrent therapy with any HMG-CoA reductase inhibitor
2. previous history of the side effects associated with any HMG-CoA reductase inhibitor
3. life-threatening arrhythmia
4. severe chronic congestive heart failure
5. hepatic dysfunction
6. renal failure
7. cerebrovascular disease
8. poor controlled diabetes
9. pregnancy, lactation
10. age <20 years
11. disability of taking medicine or absence of a written informed consent
12. Patients whom the doctors consider inappropriate by any other reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Combination of death, non-fatal myocardial infarction, unstable angina, coronary revascularization (except anticipated revascularization before randomization), non-fatal stroke and re-hospitalization due to heart failure or other cardiac causes. | 20, 50 and 80% of the projected number of patients have been enrolled in the study

SECONDARY OUTCOMES:
Each component of the primary outcome measures. | 20, 50 and 80% of the projected number of patients have been enrolled in the study

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Higashi-Osaka City General Hospital, Higashiosaka, Osaka
  - Kawachi General Hospital, Higashiosaka, Osaka
  - Osaka Minami Medical Center, National Hospital Organization, Kawachi-Nagano, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Osaka University Hospital, Suita, Osaka